CLINICAL TRIAL: NCT01456741
Title: Endobronchial Needle Aspiration With Rapid On-Site Evaluation in the Diagnosis of Central Malignant Lesions, a Randomized Controlled Trial
Brief Title: The Role of Endobronchial Needle Aspiration With Rapid On-site Evaluation in the Diagnosis of Central Malignant Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Fabiano Di Marco, M.D., Ph.D., University of Milan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: EBNA08091976
Record Dates: First submitted 2011-10-20; First posted 2011-10-21 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Lung Cancer
Keywords: endobronchial needle aspiration (EBNA); transbronchial needle aspiration (TBNA); rapid on-site evaluation (ROSE); lung cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1-EBNA with ROSE (Experimental)
  Interventions: Procedure: EBNA with ROSE
- 1-EBNA without ROSE (Experimental)
  Interventions: Procedure: standard EBNA

INTERVENTIONS:
Procedure: EBNA with ROSE — The patients in this arm will undergo:
  A) bronchoscopy, endobronchial needle aspiration (EBNA) with a cytologic needle (21 gauge), at least three forceps biopsies, bronchial brushing and bronchial washing in this procedural sequence with rapid on-site evaluation
  B) if A will be negative transthoracic needle aspiration or surgical biopsy will be performed
  C) if A and B will be negative follow-up with computed tomography or positron emission tomography and computed tomography
  Arms: 1-EBNA with ROSE
Procedure: standard EBNA — The patients in this arm will undergo:
  A) bronchoscopy, endobronchial needle aspiration (EBNA) with a cytologic needle (21 gauge), at least three forceps biopsies, bronchial brushing and bronchial washing in this procedural sequence.
  B)if A will be negative transthoracic needle aspiration or surgical biopsy will be performed
  C) if A and B will be negative follow-up with computed tomography or positron emission tomography and computed tomography
  Arms: 1-EBNA without ROSE

SUMMARY:
Endobronchial lung cancer tend to manifest in three different patterns. It can present as a bulky, exophytic mass lesion, submucosal infiltration or extrinsic compression from peribronchial disease. Bronchoscopy with differents techniques as forceps biopsy, bronchial brushing and bronchial washing is recognized as the gold standard to diagnose central airways lung neoplasms. Some authors suggested that the addition of endobronchial needle aspiration (EBNA) to these conventional diagnostic methods may increase the sensitivity of bronchoscopy in submucosal and peribronchial disease but few prospective trials have been performed and this procedure is still underutilized in many centers. Rapid on-site evaluation (ROSE) showed to improve yield of transbronchial needle aspiration (TBNA) of mediastinal nodes and pulmonary peripheral lesions, reducing the number of inadequate specimens and costs. However, its utility during endobronchial needle aspiration has not been substantiated.

This prospective study has two primary objectives: to compare the sensitivity of ROSE-EBNA with that of the conventional technique and to investigate the diagnostic yield of endobronchial needle aspiration and its contribution to CDM in the evaluation of patients with endobronchial lesions.

ELIGIBILITY:
Inclusion Criteria:

* consecutive adult patients with a suspected central lung cancer at a chest CT scan who need a bronchoscopy for diagnostic purposes

Exclusion Criteria:

* presence of uncontrolled coagulopathy, preexisting known malignancies, and the refusal to sign an informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2011-08; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
the sensitivity of the technique of endobronchial needle aspiration with rapid on-site evaluation for the diagnosis of endobronchial lung cancer | 10 day
  to determinate the sensitivity of endobronchial needle aspiration with rapid on-site evaluation compared to the conventional technique for the diagnosis of endobronchial lung cancer
the diagnostic yield of adding endobronchial needle aspiration (with and without rapid on-site evaluation) to conventional diagnostic methods for the diagnosis of endobronchial lung cancer | 10 days
  to investigate the diagnostic yield of adding endobronchial needle aspiration (with and without rapid on-site evaluation) to conventional diagnostic methods versus conventional diagnostic methods (bronchoscopy with forceps biopsies, bronchial brushing and bronchial washing) for the diagnosis of endobronchial lung cancer

SECONDARY OUTCOMES:
the impact of rapid on-site evaluation on number of passes during endobronchial needle aspiration | 30 min
  study if the presence of rapid on-site evaluation during endobronchial needle aspiration may reduce the number of passes suggested by literature

CONTACTS AND LOCATIONS:
Overall Officials: Michele Mondoni, MD, Study Director — Clinica di Malattie dell'Apparato Respiratorio, Ospedale San Paolo, Università degli Studi di Milano, Milan, Italy; Paolo Carlucci, MD, Study Chair — Clinica di Malattie dell'Apparato Respiratorio, Ospedale San Paolo, Università degli Studi di Milano, Milan, Italy; Stefano Centanni, MD, Principal Investigator — Clinica di Malattie dell'Apparato Respiratorio, Ospedale San Paolo, Università degli Studi di Milano, Milan, Italy
Locations (1):
- Clinica di Malattie dell'Apparato Respiratorio, Ospedale San Paolo, Università degli Studi di Milano, Milan, Milan, Italy